CLINICAL TRIAL: NCT00932230
Title: The Effect of Kinesio Taping on Ankle Proprioception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Principal Investigator, Dennis Enix, DC, MBA, Assistant Professor, Logan College of Chiropractic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD0206090175; 391
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Sprains and Strains
MeSH Terms: conditions — Sprains and Strains | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): An elastic tape that will be placed on subject's ankles to determine whether ankle proprioception is improved
  Interventions: Other: KinesioTape

INTERVENTIONS:
Other: KinesioTape — An elastic tape that will be placed on subject's ankles to determine whether ankle proprioception is improved

SUMMARY:
This study examines the effect of kinesiology tape on proprioception and postural control in subjects with sub-acute and chronic ankle sprains/strain.

DETAILED DESCRIPTION:
The a priori hypothesis of this study is that proprioception (knee repositioning error) and balance (sway velocity and center of pressure) will improve significantly after intervention (Kinesiotape) in participants with a history of acute or chronic ankle sprains/strains.

ELIGIBILITY:
Inclusion Criteria:

* Logan student, staff, or faculty
* Between the ages of 20 and 65
* Previous history of ankle instability/sprains
* A score of 6 out of 10 questions answered yes on the Functional Ankle Instability form will qualify the candidate

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Joint Position sense testing and postural control (sway velocity center of pressure) | Day 1, Day 2 and Day 3 of Study

SECONDARY OUTCOMES:
VAS | Day 1, Day 2 and Day 3 of Study

CONTACTS AND LOCATIONS:
Locations (1):
- Logan University, College of Chiropractic, St Louis, Missouri, United States